CLINICAL TRIAL: NCT06153758
Title: A Phase 1, 4-Part, Open-Label, Randomized Study With A 5-Period, 4 Sequence, Crossover Design to Compare the Single Dose Pharmacokinetics Between Immediate and Modified Release Formulations of Danuglipron Administered Orally to Healthy Adult Participants
Brief Title: Study to Learn How Different Forms of The Study Medicine Called Danuglipron Are Taken up Into the Blood In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C3421074
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healthy Participants; Healthy Subjects
MeSH Terms: interventions — danuglipron

STUDY DESIGN:
Intervention Model Description: 4-Part
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental): Participants will receive a single oral dose of danuglipron on Day 1 of each period
  Interventions: Drug: Danuglipron
- Part B (Experimental): Participants will receive a single oral dose of danuglipron on Day 1 of each period
  Interventions: Drug: Danuglipron
- Part C (Experimental): Participants will receive a single oral dose of danuglipron on Day 1 of each period
  Interventions: Drug: Danuglipron
- Part D (Experimental): Participants will receive a single oral dose of danuglipron on Day 1 of each period
  Interventions: Drug: Danuglipron

INTERVENTIONS:
Drug: Danuglipron — Danuglipron oral tablets
  Other Names: PF-06882961

SUMMARY:
The purpose of the study is to learn how different forms of a study medication called danuglipron are taken into the blood in healthy adults, following single dose administration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and overtly healthy
* Body mass Index (BMI) between 16-32 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria:

* Evidence or history of clinically significant medical conditions or laboratory abnormality
* Any condition possibly affecting drug absorption
* Known intolerance/hypersensitivity to a GLP-1 R agonist
* Use of prescription drugs, nonprescription drugs, dietary supplements or herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of danuglipron in each part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Parts A, C and D only: Area under the concentration-time curve from time zero extrapolated to infinite time (AUCinf), as data permit, for danuglipron in the fasted state | Predose to 48 hours post danuglipron administration
Parts A, C and D only: Maximum observed concentration (Cmax) for danuglipron in the fasted state | Predose to 48 hours post danuglipron administration
Parts A, C and D only: Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) for danuglipron (only if AUCinf is not reportable) in the fasted state | Predose to 48 hours post danuglipron administration
Part B only: Dose normalized area under the concentration-time curve from time zero extrapolated to infinite time (AUCinf,dn), as data permit, for danuglipron in the fasted state | Predose to 48 hours post danuglipron administration
Part B only: Dose normalized maximum observed concentration (Cmax,dn) for danuglipron in the fasted state | Predose to 48 hours post danuglipron administration
Part B only: Dose normalized area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast,dn) for danuglipron (only if AUCinf,dn is not reportable) in the fasted state | Predose to 48 hours post danuglipron administration

SECONDARY OUTCOMES:
All Parts: Number of Participants reporting Treatment Emergent Adverse Events | From baseline up to 28-35 days post last dose taken
All Parts: Number of Participants reporting Clinically Significant ECG Abnormalities | From baseline up to 28-35 days post last dose taken
All Parts: Number of Participants reporting Clinically Significant Vital Sign Abnormalities | From baseline up to 28-35 days post last dose taken
All Parts: Number of participants reporting clinically significant clinical laboratory abnormalities | From baseline up to 28-35 days post last dose taken
All Parts: Area under the concentration-time curve from time zero extrapolated to infinite time (AUCinf), as data permit, for danuglipron in the fed state | Predose to 48 hours post danuglipron administration
All Parts: Maximum observed concentration (Cmax) for danuglipron in the fed state | Predose to 48 hours post danuglipron administration
All Parts: Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) for danuglipron (only if AUCinf is not reportable) in the fed state | Predose to 48 hours post danuglipron administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421074